CLINICAL TRIAL: NCT03520543
Title: Positron Emission Tomography Study of alpha2-adrenergic Receptors With [11C]Yohimbine
Brief Title: [11C]Yohimbine PET Study of alpha2-AR
Acronym: [11C]Yohimbine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL17_0196; 2018-000380-82 (EudraCT Number)
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2020-02

CONDITIONS: Healthy Controls
Keywords: PET imaging; Noradrenaline; Radiotracer
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A : Imput function (Experimental): Compartmental model of the volume of distribution of [11C]Yohimbine in Brain by PET
  Interventions: Drug: [11C]Yohimbine
- Part B : validity of the measure (Experimental): Part B1 : Test Retest Variability in the distribution of [11C]Yohimbine Part B2 : Percentage of alpha2-adrenergic receptor occupancy
  Interventions: Drug: [11C]Yohimbine (Part B1) and [11C]Yohimbine + clonidine (Part B2)

INTERVENTIONS:
Drug: [11C]Yohimbine — Each subject will receive an intravenous (IV) bolus injection of [11C]Yohimbine at a dose of 370 MegaBecquerel (MBq) ± 10% with concomitant arterial blood sampling. The distribution of [11C]Yohimbine in brain will be measured by dynamic PET scans obtained from the time of injection for up to 90 minutes along with measurement of the tracer input function with arterial samples for intact tracer and metabolites to establish the total and regional compartmental kinetics of [11C]Yohimbine.
  Arms: Part A : Imput function
Drug: [11C]Yohimbine (Part B1) and [11C]Yohimbine + clonidine (Part B2) — Part B1 : Test Retest Variability will be assessed on percent difference in the binding potential following [11C]Yohimbine PET scan (IV bolus injection of [11C]Yohimbine at a dose of 370 MBq ± 10%) obtained at least 1 week after [11C]Yohimbine PET scan of part A.
  Part B2 : Occupancy of alpha2-adrenergic receptors in brain by clonidine will be evaluated by comparing the binding potential of [11C]Yohimbine (IV bolus injection of [11C]Yohimbine at a dose of 370 MBq ± 10%) after single oral dose of clonidine (0,15mg) to the binding potential of [11C]Yohimbine obtained at baseline (part A).
  Arms: Part B : validity of the measure

SUMMARY:
The main purpose of this study is to model tissue specific kinetics of [11C]Yohimbine in healthy male participants by positron emission tomography (PET) and the appropriate arterial input function (part A) ; to determine the reproducibility of measures (classical test-retest study, part B1) and to measure the blocking of [11C]Yohimbine uptake in the brain following single oral dose administration of clonidine (part B2).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Age between 20 years and 35 years
* Weight between 50kg and 90kg
* Without neurologic or psychiatric history
* Without head trauma history including loss of consciousness superior to 30 minutes.
* Affiliated to a social security or similar scheme
* Not subject to any legal protection measures
* Participant must have signed an informed consent document indicating that they understand the purpose of, and procedures required for, the study and are willing to participate in the study and comply with the study procedures and restrictions

Exclusion Criteria:

* Allen test (assessing the arterial blood flow to the hand) indicating abnormal blood supply to the hand
* Subject with orthostatic hypotension
* Subject with alcohol or substance abuses history
* Subject with somatic drug therapies
* MRI contraindications (implanted or embedded metal objects in the head or body)
* PET contraindications
* Clonidine contraindications
* Exposed to 1 millisievert or more of ionizing radiation in the year before the start of this study
* Subject unable to sign written consent for participation in the study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Binding potentials | 180 minutes
  Binding potentials are calculated using compartmental modelling techniques

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 7 days after part B
  An adverse effect is any untoward medical events that occur in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product

CONTACTS AND LOCATIONS:
Overall Officials: Chloe LAURENCIN, MD, Principal Investigator — Service de neurologie C
Locations (1):
- Service de Neurologie C - Hôpital Neurologique et Neurochirurgical Pierre Wertheimer, GHE, Bron, France

REFERENCES:
- [Result] Laurencin C, Lancelot S, Merida I, Costes N, Redoute J, Le Bars D, Boulinguez P, Ballanger B. Distribution of alpha2-Adrenergic Receptors in the Living Human Brain Using [11C]yohimbine PET. Biomolecules. 2023 May 15;13(5):843. doi: 10.3390/biom13050843. PMID 37238713